CLINICAL TRIAL: NCT04857879
Title: A Pilot Randomized Controlled Trial to Assess the Implementation and Outcomes of Good Life With Osteoarthritis (GLA:D) Program in West Virginians Suffering From the Osteoarthritis of the Knee
Brief Title: Implementation of GLA:D Program in West Virginians With Osteoarthritis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marshall University (Other)
Collaborators: University of Toronto (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Saurabh, Associate Professor, School of Physical Therapy, Marshall University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1544552
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis, Knee
Keywords: knee arthritis; Good Life with Osteoarthritis in Denmark; neuromuscular exercises
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good Life with Osteoarthritis (GLA:D) Program (Experimental): Participants will attend 2 sessions aimed at providing disease-specific education followed by 12 sessions of neuromuscular exercises, each 1 hour in length, delivered twice a week over 6 weeks.
  Interventions: Other: GLA:D program (Good Life with osteoArthritis in Denmark)
- Control intervention group (Active Comparator): Participants allocated to the control intervention will receive disease-specific education and training to learn home exercises in a 1-hour group session. They will receive a booster session 4-weeks after the first session.
  Interventions: Other: GLA:D program (Good Life with osteoArthritis in Denmark)

INTERVENTIONS:
Other: GLA:D program (Good Life with osteoArthritis in Denmark) — GLA:D includes disease-specific education combined with neuromuscular exercises. Control interventions include disease-specific education combined with exercises to optimize movement and strength of the affected knee.
  Other Names: Control intervention

SUMMARY:
This study will examine feasibility of implementing Good Life with Osteoarthritis in Denmark (GLA:D) program in West Virginians with osteoarthritis of the knee

DETAILED DESCRIPTION:
Using West Virginia (WV) as an implementation site, this study will examine the feasibility of process implementation and effectiveness of the Good Life with Osteoarthritis in Denmark (GLA:D) program in individuals with osteoarthritis of the knee (KOA). Specifically, the study will examine the feasibility and acceptability of the GLA:D program in individuals with KOA. This study will also assess the magnitude of changes in self-reported knee pain and functional impairments as well as physical performance in individuals who receive GLA:D compared to those who receive control interventions consisting of disease-specific education and exercises for KOA.

ELIGIBILITY:
Inclusion Criteria:

1. Between 45 to 90 years of age,
2. Osteoarthritis of the knee (KOA) (Kellgren and Lawrence grade 2, 3, or 4) confirmed by an orthopedic surgeon based on plain film radiographs and symptoms, and
3. Recommendation by an orthopedic surgeon to pursue conservative management of KOA.

Exclusion Criteria:

1. Prior joint replacement surgery in the ipsilateral knee,
2. Known history of cognitive impairments or any neurodegenerative disease,
3. Any other neurological or musculoskeletal pathologies that have resulted in permanent mobility deficits or functional impairments,
4. Medical conditions that would preclude them from participating in exercise programs, and
5. Inability to read and comprehend English.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score (KOOS4) scores from baseline to 12-weeks later | 12-weeks
  The KOOS4 is a variant of full length KOOS that has all subscales of full length KOOS (pain, symptoms, ADL, and QOL) except sports and recreation activities subscale. There are 9 items in the pain subscale, 7 items in the symptom subscale, 17 items in the ADL subscale, and 4 items in the QOL subscale. The items across these subscales are scored on the scale of 0 to 4 where 0 indicates no problem and 4 indicates an extreme problem. Each subscale has sufficient stability and dimensionality, and therefore the score for each subscale is calculated independently on 0-100 interval with 0 indicating an extreme problem and 100 indicating no problems.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Therapy, Marshall University, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No